CLINICAL TRIAL: NCT06701227
Title: In Situ Simulation in Prenatal Breastfeeding Education
Brief Title: Breastfeeding Simulation in Prenatal Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Taison Regis Penariol Natarelli, PhD student, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4.324.588
Record Dates: First submitted 2024-11-18; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Breastfeeding Self-Efficacy; Exclusive Breastfeeding
Keywords: Breast Feeding; Simulation Training; Health Education; Prenatal Education
MeSH Terms: conditions — Breast Feeding; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In Situ Simulation (Experimental): The educational intervention consists of applying the in situ simulation scenario entitled "Breastfeeding the Newborn", previously structured and validated among experts, through individual home visits, with pregnant people.
  Interventions: Other: In Situ Simulation
- Routine Prenatal Care (No Intervention): Routine prenatal guidance on breastfeeding. Currently, prenatal education provided by the Unified Health System (UHS) is being carried out through individual counseling during prenatal consultations and in groups for pregnant people organized by the FHUs and also by the local maternity hospital.

INTERVENTIONS:
Other: In Situ Simulation — The simulation scenario included briefing (5 min), scenario (10 min), and debriefing (20 min).
  Materials and Simulators: neonatal mannequin, with its crying controlled by a smartphone; breastfeeding simulator that had the function of ejecting liquid imitating human milk.
  Team: One facilitator and one actor playing a Community Health Worker.
  Arms: In Situ Simulation

SUMMARY:
Breastfeeding education should be initiated during pregnancy. Simulation is an effective educational technique that has been little explored in the context of prenatal education.

This study aims to evaluate the feasibility and effectiveness of an in situ simulation scenario about breastfeeding, as a prenatal educational intervention at home, on breastfeeding self-efficacy and related outcomes.

DETAILED DESCRIPTION:
According to the World Health Organization, breastfeeding should be initiated within the first hour of life, being exclusive for children up to six months of age, complemented and continued for up to two years or more. However, despite the countless benefits of human milk for both maternal and child health and for society as a whole, establishing and maintaining breastfeeding, in accordance with international guidelines, is still a challenge. Low breastfeeding rates can be observed in several countries around the world.

Breastfeeding education should be initiated during prenatal care. Studies indicate that high quality education throughout prenatal care is a protective factor for the success of breastfeeding. However, pregnant people are not always properly advised about breastfeeding. Most of the times, breastfeeding education in prenatal care is carried out through traditional teaching methods, which are more based on behavioral education and do not encourage an individual's autonomy in the teaching-learning process.

On the other hand, experiential learning is more related to constructive education, by encouraging the co-creation of a learning environment, where the teacher/nurse becomes a facilitator based on the learner's needs. Clinical simulation is an educational technique that promotes an active learning experience, through the imitation of reality in a safe and controlled environment, being able to increase participant's knowledge, skills, confidence, and clinical judgment. Among the existing simulation modalities, in situ simulation stands out as the one that takes place in the real environment (hospitals, outpatient clinics, and community). In situ simulation has several specific advantages from an educational and economic point of view.

Simulation has already been used in breastfeeding teaching. Some studies describe and evaluate the use of simulation-based education to teach breastfeeding to undergraduate and postgraduate students, as well as for lactation support providers training. Multiple types of simulation have been used to teach breastfeeding, including hybrid simulation, Objective Structured Clinical Examination, telesimulation and virtual simulation.

However, there is little literature exploring the use of simulation for the education of patients. Usually, experiences using simulators to teach pregnant and postpartum people about breastfeeding do not consist of structured and validated scenarios, focusing only on demonstrating the breastfeeding technique with low-fidelity simulators. There are no studies in the literature about in situ simulation scenarios created specifically for patients and implemented in the community.

Based on Bandura's theory of self-efficacy, first, it is necessary for pregnant people to believe that they are capable of breastfeeding and then seek resources, internal or external, to assist them in this practice. The following sources of information support breastfeeding self-efficacy: personal experience; observational or vicarious experience; verbal persuasion and emotional and physiological state, with personal experience considered the main source of information for self-efficacy. Therefore, a simulation scenario could be able to promote a personal breastfeeding experience for pregnant people, although simulated, yet highly realistic.

Therefore, this study aims to evaluate the feasibility and effectiveness of an in situ simulation scenario about breastfeeding, previously created and validated with experts, specifically for pregnant people, as a prenatal educational intervention at home, on breastfeeding self-efficacy and related outcomes (exclusive breastfeeding rate and breastfeeding related difficulties at 2 months after childbirth).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant people registered at a FHU in the city in their third trimester of pregnancy.

Exclusion Criteria:

* Present with a pre-existing health condition that constitutes a permanent contraindication for breastfeeding (people infected with HIV, HTLV1, or HTLV2).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Change of breastfeeding self-efficacy measured by applications of the Brazilian-Portuguese version of the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) from baseline to 2 months after delivery | At baseline (pre-test), immediately after educational intervention/in situ simulation (immediate post-test) and 2 months after childbirth (follow-up post-test)
  The BSES-SF is a scale consisting of 14 items, using a 5-point Likert scale, that measures a person's self-confidence in their abilities to breastfeed. The total score can range from 14 to 70 points, with 14 representing the lowest level of self-efficacy and 70 the highest possible, further divided into: low efficacy (14-32 points), medium efficacy (33-51 points), and high efficacy (52-70 points) (Dennis, 2003). The results will be presented as the mean scores of the BSES-SF, which will be statistically analyzed and compared
Exclusive breastfeeding rate (number of babies who are being fed exclusively with breast milk, and no other liquids or solids, except in specific cases such as vitamins, mineral supplements, or medications) by a self-developed questionnaire | At 2 months after delivery
  The self-developed questionnaire was reviewed by 2 experts in clinical simulation and breastfeeding, and it was administered by the principal investigator to the study participants
Breastfeeding difficulties (number of lactating people who faced difficulties such as nipple trauma, breast engorgement, mastitis, breast abscess, low milk production, ineffective sucking and others) by a self-developed questionnaire | At 2 months after delivery
  The self-developed questionnaire was reviewed by 2 experts in clinical simulation and breastfeeding, and it was administered by the principal investigator to the study participants

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Mara Monti Fonseca, RN, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Municipal Health Department, Jaboticabal, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No